CLINICAL TRIAL: NCT06499337
Title: Evaluation of the Feasabilty and Acceptability of a Safety Plan After Suicidal Attempt to Prevent Recurrence After an Emergency Department Admission.
Brief Title: Safety Plan in Emergency Department to Prevent Suicidal Attempt Recidive
Acronym: PLUS
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D21_PEPI-0011
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Suicidal Ideations; Suicidal Attempt; Prevention; Safety Plan
Keywords: Safety plan; Suicidal attempt; feasability; acceptability
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Suicide is one of the leading causes of death worldwide, with more than 700 000 deaths due to suicide every year, according to the World Health Organisation (WHO). In France, mortality rate by suicide is 17% higher than the European average; moreover, around 7% if the population (aged 18-75 years old) attempted suicide in their life.

Since years 2000, a series of preventative interventions have been developed to reduce suicide risk, with perhaps the most widely used is suicide safety planning. Several studies showed positive results after evaluating the efficacy of suicide safety planning for reducing patient risk. However, this intervention hasn't been yet evaluated in French emergency department settings.

Safety planning is a collaborative intervention between a therapist and the patient, by which a series of preventive actions are planned in the event patient experiences suicide ideation. Patients are provided with a paper form of the completed safety plan, including the following: personal warning signs, self-management strategies, reasons for living, social supports, and crisis supports.

In this study, we aim to assess the feasability and the acceptabilty of using the safety plan among patients hospitalised in a short-term unit, after an emergency department admission for suicidal attempt.

DETAILED DESCRIPTION:
Suicide is one of the leading causes of death worldwide, with more than 700 000 deaths due to suicide every year, according to the World Health Organisation (WHO). In France, mortality rate by suicide is 17% higher than the European average; moreover, around 7% if the population (aged 18-75 years old) attempted suicide in their life.

Since years 2000, a series of preventative interventions have been developed to reduce suicide risk, with perhaps the most widely used is suicide safety planning, which is a brief intervention to help individuals who survived a suicide attempt to develop a set of tools and steps, to reduce the likelihood of engaging in suicidal behaviour. Several studies showed positive results after evaluating the efficacy of suicide safety planning for reducing patient risk. Recently, a systematic review concluded that Safety Planning is a valuable intervention for patients experiencing suicide-related distress, and was associated with improvements in suicidal ideation and behaviour and reductions in hospitalizations. Qualitative studies suggest a Safety Planning intervention is acceptable and feasible, as well as adaptable to the clinical area in its modality and delivery. Despite positive outcomes, this intervention has not been fully evaluated in French settings. A previous study concluded it was not adapted to emergency department due to a lack of time or available exam rooms for professionals to conduct the intervention. Therefore, in our study, participants will be recruited in a post-ED unit, where patients are monitored for maximum 72 hours, before being discharged home or transferred to hospital facilities.

Safety planning is a collaborative intervention between a healthcare worker and the patient, by which a series of preventive actions are planned in the event patient experiences suicide ideation. Safety planning included identifying: 1) warning signs or triggers that indicate suicide ideation is likely to occur, 2) internal coping strategies (e.g., distracting activities) for use when those triggers occur or when experiencing suicide ideation, 3) social contacts for further distraction or social locations that may provide distraction, 4) supportive contacts (who can provide assistance), 5) emergency resources (e.g., therapist phone numbers, hotlines, local hospital emergency room locations), and also included steps to ensure the safety of the home environment that minimize the patient's ability to act on suicidal thoughts or urges (i.e., reducing access to lethal means).

In this study, Safety plan was delivered face-to-face, during the post-ED stay; upon discharge, participants were provided with the paper-based plan they completed with their physician.

The main outcome of our study was to evaluate the feasibility - assessed by healthcare workers- and the acceptability - from patients' point of view- of conducting a Safety plan in a post-ED setting, after suicidal attempt. Secondary outcomes included to evaluate Safety plan utility, assessed by patients based on their use or not of the Safety plan at 1 and 6 months after inclusion, and its efficacy, on the recurrence of suicidal attempt over the 6 months after inclusion.

To evaluate the outcomes at 1 and 6 months, patients were recontacted by a psychologist to complete a brief questionnaire over the phone.

At baseline, we also collected sociodemographics information, including marital status and living situation; patients completed the Hospital anxiety and depression scale, and suicidal ideations evaluated with the Columbia-Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patients hospitalised in a post-emergency unit following a suicidal attempt

Exclusion Criteria:

* Patients whose clinical state or French level prevent to understand the information regarding the study and to consent to the study
* Pattients whose clinical state or French level prevent to participate to the Safety plan intervention
* patients who do not agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals included in the study were patients hospitalized at the post-emergency short-term psychiatric unit following a visit to the emergency room for a suicide attempt. The recruitment took place between June 2022 and December 2023. Patients eligible for inclusion had to be adults, admitted to the hospital following a suicide attempt, and willing to participate in the study. The criteria for non-inclusion were: a) patients who were minors, b) patients who were unable to be informed or to understand the course of the study (if they did not understand French or if their condition did not allow it), c) patients who were opposed to the collection of data for research purposes, d) patients whose psychiatric and/or somatic condition was incompatible with the brief intervention and/or the study questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Day of intervention (D0)
  The feasibility of implementing the safety plan was assessed with a questionnaire submitted to the caregivers who delivered the intervention. This self-administered questionnaire assessed: the time required to complete the safety plan, the availability of a suitable location for conducting the interview, the clinical and mood status of the individuals, and the difficulties encountered during the intervention. This questionnaire determined the feasibility score ranging from -4 to 6.
Acceptability | Day of intervention (D0)
  A questionnaire for patients who had benefited from the safety plan was used to establish an overall acceptability score intervention. This questionnaire, partly based on Stanley's evaluation, allowed to determine an acceptability score, ranging from -8 to 8, a high positive value indicating a higher acceptance of the intervention by the patient. The acceptability score was calculated by summing the responses to the following questions: a) Have you ever had the opportunity to participate in an interview of this type (security plan)? b) Were the questions clear? c) Were there any questions that made you uncomfortable? d) Did you find this interview lengthy? e) Did you find the questions repetitive? f) Do you think you learned anything about yourself from this interview? g) Do you think the security plan can help you in your situation? h) Do you think this document could be useful to you in the future?

SECONDARY OUTCOMES:
Utility | 1 month after discharge
  Utility of the Saftey plan was assessed at 1 month, by asking participants if they retain their physical safety plan, they had use it since being discharged, and whether they find it useful.
Efficacy | Any suicidal attempt occuring up to 6 months after inclusion
  Efficacy was evaluated based on suicidal attempt recurrence over the 6 months following the intervention. Patients (or their emergency contact) were contacted by a mental healthcare worker to assess any new attempt.

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris Psychiatrie et Neurosciences, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Ganay M, Duroy D, Perozziello A, Lejoyeux M, Geoffroy PA. Study assessing the feasibility and acceptability of implementing the Safety Plan for suicide prevention in a French emergency department. Encephale. 2023 Dec;49(6):656-657. doi: 10.1016/j.encep.2023.03.002. Epub 2023 Apr 28. No abstract available. PMID 37121806